CLINICAL TRIAL: NCT01521936
Title: Vitamin D3 Supplementation in Acute Myeloid Leukemia: Pharmacokinetic Study
Brief Title: Cholecalciferol in Treating Patients With Acute Myeloid Leukemia Undergoing Intensive Induction Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 201311; NCI-2011-03554 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (25(OH)-D3 levels 20-31.9 ng/mL [insufficient levels]) (Experimental): Patients receive a loading dose of cholecalciferol PO on day 1. Patients then receive lower-dose cholecalciferol PO beginning on day 8.
  Interventions: Dietary Supplement: cholecalciferol; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (25(OH)-D3 levels 20-31.9 ng/mL [insufficient levels]) (Experimental): Patients receive a loading dose of cholecalciferol PO on day 1. Patients then receive higher-dose cholecalciferol PO beginning on day 8.
  Interventions: Other: pharmacological study; Dietary Supplement: cholecalciferol; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given PO (lower dose)
  Other Names: Calciol; Vitamin D3
  Arms: Arm I (25(OH)-D3 levels 20-31.9 ng/mL [insufficient levels])
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Dietary Supplement: cholecalciferol — Given PO (higher dose)
  Other Names: Calciol; Vitamin D3
  Arms: Arm II (25(OH)-D3 levels 20-31.9 ng/mL [insufficient levels])
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This partially randomized phase II trial studies the side effects and best way to give and best dose of cholecalciferol in treating patients with acute myeloid leukemia (AML) undergoing intensive induction chemotherapy. Cholecalciferol may help improve the outcome of patients with AML undergoing intensive chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess patients with regards to changes in 25(OH)-D3 changes after supplementation. II. To develop a pharmacokinetic model to describe the time course of the relationship of vitamin D3 (cholecalciferol) supplementation that drives the levels of 25(OH)-D3 during the intensive induction chemotherapy. III. To determine the safety and toxicity of vitamin D3 supplementation in AML patients undergoing intensive induction chemotherapy. SECONDARY OBJECTIVES: I. To explore whether rapid (loading dose of vitamin D3) normalization of 25(OH)-D3 levels will have an effect on the progression free and overall survival. II. To explore whether a relationship exists between the pharmacokinetics of the 25-hydroxy-vitamin D3 and white blood cell count. OUTLINE: Patients with pretreatment 25(OH)-D3 levels 20-31.9 ng/mL (insufficient levels) are randomized to 1 of 2 treatment arms. ARM I: Patients receive a loading dose of cholecalciferol orally (PO) on day 1. Patients then receive lower-dose cholecalciferol PO beginning on day 8. ARM II: Patients receive a loading dose of cholecalciferol PO on day 1. Patients then receive higher-dose cholecalciferol PO beginning on day 8. Patients with pretreatment 25(OH)-D3 levels < 20 ng/mL (deficient levels) receive a loading dose of cholecalciferol PO on days 1 and 8. Patients then receive lower-dose cholecalciferol PO beginning on day 15. For all patients, treatment continues in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria: Pathologic diagnosis of newly diagnosed AML (excluding acute promyelocytic leukemia [APL]) Patients undergoing intensive induction therapy (equivalent of 7+3, cytarabine, daunorubicin, etoposide [ADE] or high-dose cytarabine containing regimens) Subnormal 25(OH)-D3 levels (< 32 ng/mL) Serum calcium =< upper limit of normal Demonstrate the ability to swallow and retain oral medication Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure Exclusion Criteria: Patients should not have a history of nephrocalcinosis Patients should not have received bisphosphonate treatment within 28 days before study entry Pregnant or nursing female patients Unwilling or unable to follow protocol requirements Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug Received an investigational agent within 30 days prior to enrollment Patients who cannot be discontinued from cimetidine, thiazide diuretics and/or heparin Patients who are on magnesium based antacids who cannot be offered an alternative regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in 25(OH)-D3 levels after supplementation | From baseline to monthly for the first 3 months and then every 3 months
  The within-group pre- and post-supplementation levels will be summarized separately and the within-subject change will also be computed. To assess within-arm treatment effects the sign test will be used.
Pharmacokinetic parameters | 30 minutes before administration, 30 minutes after administration, and 24 hours after administration on day 1; monthly for the first 3 months; and then every 3 months
  Summarized using the mean (with corresponding 90% confidence intervals) and standard deviation.
Safety and toxicity parameters | Daily for 21 days and monthly thereafter, up to 30 days after last dose of study drug
  Rates corresponding to toxicity endpoints will be estimated using simple relative frequencies. The corresponding 90% confidence intervals for the estimated probabilities will be computed using the method proposed in Clopper and Pearson. Comparison between groups will be done in an exploratory fashion using appropriate two-sample tests. A nominal significance level of 0.10 will be used in all testing.

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States